CLINICAL TRIAL: NCT07316972
Title: CEST-based Biomarkers to Delineate the Epileptogenic Zone
Acronym: CEST-BEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MQS_2024_10
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy (Treatment Refractory)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients scheduled to undergo a pre-surgical evaluation for drug-resistant epilepsy. (Experimental)
  Interventions: Other: CEST sequence on a 7-Tesla MRI

INTERVENTIONS:
Other: CEST sequence on a 7-Tesla MRI — CEST sequence on a 7-Tesla MRI

SUMMARY:
Epilepsy is a common neurological disorder with an incidence of 1%. Although many anti-seizure medications are available, about 30% of patients are resistant to drug treatments. Epilepsy surgery is an effective treatment for some of these patients. It involves removing the brain region responsible for generating seizures, called the epileptogenic zone (EZ).

A pre-surgical evaluation is performed to locate and delineate the region where seizures originate (the seizure onset zone [SOZ]) and to confirm that this zone is unique and accessible for surgery-that is, that the potential benefits outweigh the risks of functional deficits resulting from its removal. The lesion itself is identified and characterized through post-operative histological examination and, in some cases, based on MRI criteria.

During pre-surgical evaluation, in cases where no lesion is visible on MRI or when surface EEG suggests that a large or multiple epileptic networks may be involved, stereo-electroencephalography (SEEG) is the method of choice to delineate the area for resection. However, SEEG has limitations: it is invasive and records from a restricted brain volume.

Despite advances in neuroimaging techniques, the localization of the epileptogenic zone and mapping of functional brain alterations still need improvement beyond what morphological MRI anomalies can reveal.

Because epileptic tissue is characterized by increased neuronal excitability and metabolic abnormalities, techniques that allow precise evaluation of these changes could deepen our understanding of the disease and provide new tools for epilepsy surgery. An alternative MRI approach based on metabolite quantification using chemical exchange saturation transfer (CEST) has been suggested to aid in localizing the epileptogenic zone in preliminary studies. However, limited availability of ultra-high-field MRI, low localization precision of the epileptogenic zone, and lack of systematic validation in patients have delayed its clinical use.

This study aims to explore a cohort of patients with temporal lobe epilepsy who are candidates for surgery using CEST MRI. We will quantify glutamate and glucose concentrations using glu-CEST and gluco-CEST, respectively, and correlate the results with the localization of the epileptogenic zone determined by pre-surgical evaluation, and where applicable, SEEG and post-operative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with drug-resistant temporal lobe epilepsy (mesial or lateral)
* Requiring a pre-surgical evaluation including long-term video EEG
* At least 5 of them will be recruited after surface video EEG indicates the need for further exploration by SEEG
* With or without a radiologically visible lesion

Exclusion Criteria:

* Absolute or relative contraindication to MRI (metallic implants, including intrauterine devices other than the MIRENA® brand, claustrophobia, etc.)
* Expected inability to remain still for 90 minutes in a 7T MRI
* Diabetic individuals
* Individuals under legal protection measures
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Glucose concentration measured by CEST in the the seizure onset zone (SOZ) | Day 0

SECONDARY OUTCOMES:
Glucose concentration measured by CEST in the irritative zone (IZ) | Day 0
Glucose concentration measured by CEST in the propagation zone | Day 0
Glutamate concentration measured by CEST in the seizure onset zone (SOZ) | Day 0
Glutamate concentration measured by CEST in the irritative zone (IZ) | Day 0
Glutamate concentration measured by CEST in the propagation zone | Day 0